CLINICAL TRIAL: NCT03285399
Title: Micronutrient Status in Breastfeeding Women and Their Children in Bhaktapur Nepal
Brief Title: Bhaktapur Maternal and Child Micronutrient Study
Status: Completed | Type: Observational
Sponsor: Centre For International Health (Other)
Collaborators: Tribhuvan University, Nepal (Other); Harvard School of Public Health (HSPH) (Other); Oslo and Akershus University of Applied Sciences (Unknown)
Responsible Party: Sponsor
Other Study IDs: 172226
Record Dates: First submitted 2017-09-13; First posted 2017-09-18 (Actual); Last update posted 2017-09-18 (Actual); Status verified 2017-09

CONDITIONS: Malnutrition, Infant; Malnutrition; Anemia
Keywords: Nepal; Breastfeeding; Micronutrients; Women; Infants
MeSH Terms: conditions — Infant Nutrition Disorders; Malnutrition; Anemia; Breast Feeding

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Breastmilk Plasma Red blood cells Urine
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Between February 2008 and February 2009, 500 infant-mother pairs in Bhaktapur, Nepal were randomly selected in this nutritional survey. The dietary intake, nutritional status of several nutrients, growth, and breastfeeding habits were measured in both the women and their infants.The objective of this first phase was to estimate the intake and status of several nutrients in relation to breastfeeding. These mother-child pairs were revisited around the child's fifth birthday when growth, diet, and neurodevelopment was measured. The objective of this phase was to create a cohort study where factors in infancy could be related with health outcomes and development 5 years later.

DETAILED DESCRIPTION:
Over a period of one year, a total of 500 lactating (encompassing both exclusive and partial breastfeeding) women were enrolled in the study and completed the first 24-hour dietary recall. The women attended a hospital for physical examination, dietary interview, and blood sampling. Blood samples were also collected from their infants who also went through a detailed clinical examination

The blood samples from mothers and infant pairs were collected approximately one week apart. The blood was spun down, plasma separated and transferred into storage vials immediately. Plasma and blood pellets were stored in cryovials at -70 until analysis.

All women were also requested to provide one breast milk and one urine sample.

Plasma, blood pellet, urine, and breast milk was stored at -70 degrees celcius until analysis.

Plasma was analyzed for iron, transferrin receptor, ferritin, cobalamin, folate, vitamin A, vitamin D, vitamin E, several amino acids and other micronutrient related metabolites.

The breast milk will be analyzed for iodine, fatty acids, and several B vitamins

The urine was analyzed for iodine.

In phase 2, after 5 years we revisited the mother-child pairs and measured growth, diet, food security, and neurodevelopment.

ELIGIBILITY:
Inclusion Criteria:

* availability of consent
* no ongoing illness
* resides in the selected cluster
* that household information could be obtained
* that the mother was lactating

Exclusion Criteria:

* refused blood sampling
* chronic illness

Ages: 2 Months to 11 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: A cross-sectional survey was carried out and 500 healthy lactating women (17-44 years old) were randomly selected from Bhaktapur municipality, Nepal. Bhaktapur is an urban area located 15 km east of the capital Kathmandu and was chosen because of the diversity of this population spanning all socio-economic strata, providing a unique opportunity to explore dietary variation.
Sampling Method: Probability Sample
Enrollment: 1000 (Actual)
Dates: Start 2008-01-12 (Actual); Primary Completion 2010-02-28 (Actual); Study Completion 2014-02-28 (Actual)

PRIMARY OUTCOMES:
Prevalence of micronutrient deficiency | 1 year
  The status and prevalence of deficiencies of several micronutrients has been estimated
Predictors for micronutrient status | 1 year
  We will estimate predictors for several of the measured micronutrients using other biomarkers and clinical and demographic variables.
Prevalence of anaemia in mothers and children | 1 year
  Hemoglobin concentration is measured for all participants and the proportion anaemic and predictors for anaemia will be presented.

SECONDARY OUTCOMES:
Neurodevelopment at 5 years | 5 years
  Neurodevelopment is measured when the children are 5 using the Ages and Stages questionnaire and the NEPSY II tests. These measures will be related to micronutrient status, inflammation and stress markers.
Growth during infancy and at 5 years of age | 5 years
  Growth (length and weight) is measured when the children are 5 years and will be related to nutritional status.
Markers of stress and inflammation. | 1 year
  Maternal and infants markers of inflammation (CRP, neopterine, kynurenic acid, kynurenine, tryphtophane, etc) and stress (leucocyte telomere length) will be measured and related to micronutrient status.
Breastmilk b-vitamin concentration | 1 year
  The concentration of several b-vitamins will be estimated in the breast milk and related to dietary intake and maternal and child status

CONTACTS AND LOCATIONS:
Overall Officials: Tor A Strand, MD/PhD, Principal Investigator — University of Bergen
Locations (1):
- Siddhi Memorial Hospital (SMH),Bhelukhel, Bhimsensthan, Bhaktapur, Nepal

IPD SHARING:
Plan to Share IPD: Undecided
Data can be requested by contacting the principal investigator (Tor Strand) or one of the other investigators.